CLINICAL TRIAL: NCT01717937
Title: Comparison of Phase-variance Optical Coherence Tomography and Fluorescein Angiography in the Imaging of Retinovascular Disease
Brief Title: Comparison of Phase-variance Optical Coherence Tomography and Fluorescein Angiography in Retinovascular Imaging
Acronym: PVOCT
Status: Terminated | Type: Observational
Why Stopped: insufficient enrollment
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: PVOCT-12-10060
Record Dates: First submitted 2012-10-28; First posted 2012-10-31 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Age-related Macular Degeneration; Diabetic Retinopathy; Hypertensive Retinopathy; Retinal Vein Occlusion; Retinal Artery Occlusion
Keywords: retinovascular disease; imaging; fluorescein angiography; FA; angiography; optical coherence tomography; OCT; phase variance; comparison; age-related macular degeneration; diabetic retinopathy; hypertensive retinopathy; retinal vein occlusion; retinal artery occlusion
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Hypertensive Retinopathy; Retinal Vein Occlusion; Retinal Artery Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PVOCT: Subjects will receive fluorescein angiography (FA) as part of their normal clinical evaluation and will undergo phase variance optical coherence tomography (PV-OCT) as the study intervention. This involves having subjects undergo standard, noninvasive optical coherence tomography (OCT) scans with an FDA-approved OCT device, and the data gathered by this device will be transferred to a separate computer for processing using novel software. This software is capable of utilizing the existing data to generate phase variance OCT images.
  Interventions: Procedure: Phase variance optical coherence tomography (PV-OCT)

INTERVENTIONS:
Procedure: Phase variance optical coherence tomography (PV-OCT) — Subjects will undergo standard, noninvasive optical coherence tomography (OCT) scans with an FDA-approved OCT device, and the data gathered by this device will be transferred to a separate computer for processing using novel software. This software is capable of utilizing the existing data to generate phase variance OCT images. There are no known risks associated with OCT scans.

SUMMARY:
The purpose of this study is to determine whether phase variance optical coherence tomography (PV-OCT), a software-based optical coherence tomography(OCT) image processing technology, can be used to generate angiographic images of the retinochoroidal vasculature that are comparable to those produced by fluorescein angiography (FA), the current gold standard diagnostic test.

DETAILED DESCRIPTION:
Fluorescein angiography (FA) has long been the gold standard for vascular imaging of the retina and choroid. It is a test that involves the intravenous injection of fluorescein dye, followed by imaging of the dye's passage through the blood vessels inside the eye. It is commonly used to diagnose many forms of retinovascular disease, as well as to assess the retina's response to various therapeutic interventions. While FA is a relatively safe diagnostic test, it carries the risk of both minor and major side effects. These include nausea and vomiting, yellowing of the skin and urine, vascular extravasation with skin eruption and necrosis, vasovagal reactions, myocardial infarction, respiratory failure, anaphylaxis, cardiopulmonary arrest, and death. Additionally, the test is time-consuming, technically difficult to perform, and requires patients to undergo the discomfort associated with intravenous access. Despite these drawbacks, FA is still commonly used in clinical practice, as there are no existing alternative tests with the ability to provide comparable detail of the retinal and choroidal vasculature.

Phase-variance optical coherence tomography is a novel, noninvasive, software-based technology capable of generating angiographic images from the data gathered by standard OCT scans. Preliminary research suggests it can produce high-definition representations of the retinal and choroidal vasculature which may be more detailed than the images produced by FA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected or established retinovascular disease who are going to undergo FA as part of their usual clinical evaluation.
2. Patients must be age 13 or above.
3. Patients must be able to speak and understand the English language in order to provide informed consent.

Exclusion Criteria:

1. Any patients who are unwilling to participate or provide informed consent.
2. Any patients who are pregnant at the time of enrollment.
3. Any patients with ocular media opacities which prevent clear evaluation of the fundus by either FA or OCT.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients seen in the University of California, San Francisco Retina Clinic with suspected or established retinovascular disease and who are scheduled to undergo fluorescein angiography as part of their normal clinical evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Measurement of to be determined physical characteristics of retinovascular structures seen on phase variance optical coherence tomography (PV-OCT) and fluorescein angiography(FA). | On the day in which a patient receives PV-OCT and FA imaging, estimated to take 2 hours.
  Masked examiners (retina specialists) will evaluate and grade coded PV-OCT and FA images for the presence and features of various retinovascular abnormalities (e.g., choroidal neovascular membranes, microaneurysms, venous dilation, etc.). Metrics to determined and may include: size, depth, area, volume, and relative position. Each subject's graded PV-OCT images will be compared to their graded FA images.

SECONDARY OUTCOMES:
Changes over time in the to be determined measured physical characteristics of retinovascular structures seen on PV-OCT and FA. | Up to 12 months after enrollment.
  Each time a subject is determined to require OCT imaging as part of their normal clinical evaluation over the duration of the study, a PV-OCT scan will also be performed. Measured to be determined physical characteristics of these scans will be compared to measurements obtained from prior PV-OCT images in order to assess changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M McClintic, M.D., Principal Investigator — University of California, San Francisco; Daniel M Schwartz, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- See also: Phase-contrast OCT imaging of transverse flows in the mouse retina and choroid. — http://www.ncbi.nlm.nih.gov/pubmed/18566457
- See also: Noninvasive imaging of the foveal avascular zone with high-speed, phase-variance optical coherence tomography. — http://www.ncbi.nlm.nih.gov/pubmed/22125275
- See also: In vivo volumetric imaging of human retinal circulation with phase-variance optical coherence tomography. — http://www.ncbi.nlm.nih.gov/pubmed/21698014